# Head and Neck Cancer Clinical Trials: Analysis of Participation Trends Among Head and Neck Cancer Patients in Clinical Trials

# An Informed Consent Form For Power Clinical Trial's Observational Clinical Study

Date: March 24, 2023

### Introduction and Key Details

The purpose of this brief summary is to provide you with an overview of our observational clinical study, focusing on the procedures, potential risks, and benefits of participation. Before you decide whether to participate, we want to remind you that your consent is required, but you are under no obligation to take part. You have the right to withdraw at any time without consequences.

Our study seeks to understand the reasons why patients with head and neck cancer choose to enroll, remain, or withdraw from clinical trials. The primary procedures involved in this study are completing questionnaires and follow-up calls. These procedures have been designed to minimize any potential risks to participants.

As an observational study, there may not be any direct medical benefits to participants. However, the data collected can be used to identify ways to improve clinical trial participation rates, ultimately benefiting patients with head and neck cancer.

The findings of this study will provide valuable insights into the factors that influence clinical trial participation rates.

By identifying these factors, we hope to improve recruitment strategies and patient engagement in clinical trials, leading to better treatment options and outcomes for head and neck cancer patients. However, it is important to emphasize that participation in this

study is voluntary. Declining to participate will not affect your rights or privileges in any way.

We strongly encourage you to review the consent form carefully and ask any questions you may have before making a decision about participation. You may also wish to discuss the study with your family, friends, trusted advisors, and healthcare professionals to ensure that you have all the information you need to make an informed decision.

Remember that your participation is entirely voluntary, and you have the right to withdraw at any time without consequences.

### The Clinical Trial's Objective

Clinical trials play a vital role in the development of new treatments for head and neck cancer. However, it is not always clear whether the participants in these studies accurately represent the larger population. Therefore, this clinical trial aims to examine the various factors that influence a patient's decision to enroll, discontinue, or resume participation in a head and neck cancer clinical trial. By understanding the factors that affect clinical trial participation rates, we can ultimately improve the effectiveness and relevance of future studies.

To ensure that the study's findings are statistically significant, we are seeking to recruit individuals from a diverse range of demographic groups. This will enable us to investigate how various factors, such as age, race, income, and education level, affect a patient's decision to participate in a clinical trial. By gathering this information, we hope to develop better strategies to increase participation rates among underrepresented groups in future clinical trials.

It is important to note that participation in this clinical trial is voluntary, and individuals have the right to withdraw at any time without consequence. The primary procedures of this observational clinical study involve answering questionnaires and making follow-up calls, with minimal risk to the participants. Nonetheless, we strongly encourage potential participants to carefully review the consent form and ask any questions they may have before deciding to participate.

Overall, this clinical trial seeks to advance our understanding of the factors that influence clinical trial participation rates among head and neck cancer patients. By

improving participation rates, we can ultimately accelerate the development of new and effective treatments for this devastating disease.

#### The Clinical Trial Procedure

We are conducting an observational clinical research study focused on understanding the factors that affect head and neck cancer patient participation in clinical trials, including reasons for enrollment, withdrawal, and completion.

Our study aims to recruit participants who are currently receiving treatment in an interventional trial, as well as those who have previously taken part in or withdrawn from a clinical trial. We will utilize electronic medical record systems to identify potential participants and invite them to participate in our study.

If you decide to participate, our staff will provide you with a consent form and explain the study's objectives and your rights as a participant. We will collect data from participants every two weeks through questionnaires that cover their demographics, medical history, and the factors that led them to enroll in, withdraw from, or complete the clinical trial. Additionally, the research team will conduct phone or video interviews with participants every three months to gather more detailed information.

The data collected will be analyzed to identify the variables that influence patient participation in clinical trials, using statistical analysis. The results of the study will be disseminated through conference presentations and scholarly journal publications, with the aim of benefiting clinical trial stakeholders.

By improving patient recruitment and retention, our findings will enhance future clinical studies for head and neck cancer patients.

It's important to note that participation in our study is entirely voluntary, and individuals have the right to withdraw at any time without any consequences. Our study procedures involve minimal risks to participants, primarily consisting of answering questionnaires and participating in follow-up interviews. If you have any questions or concerns, please do not hesitate to contact our research team

Are There Any Dangers Involved?

While observational clinical research studies for head and neck cancer do not involve experimental interventions, there may still be risks associated with participation. These risks could include potential breaches of privacy, emotional distress related to the study's topic, and negative outcomes from any procedures performed during the trial.

Before deciding to participate in the study, it is essential to carefully read and understand the informed consent form and discuss any concerns with the research team. The team will provide detailed information on the potential risks and benefits of participating in the study, as well as the measures they will take to protect participants' safety and well-being.

# Does It Have Any Benefits?

Observational clinical trials offer head and neck cancer patients a chance to contribute to the advancement of medical knowledge and potentially enhance future treatment options. Although experimental therapies are not part of these trials, patients may still receive expert care and attention during the study.

Before deciding to participate in a clinical trial, it is crucial for patients to carefully assess the potential benefits and risks based on their individual situation and objectives. It is recommended that patients discuss their options with their healthcare provider and the research team before making a decision.

# Factors That May Result in the Termination of Your Participation

It's important to understand that your participation in a clinical trial can be terminated without your consent by the researcher or sponsor for various reasons. This may include the suspension or termination of the study, the removal, suspension, or withdrawal of funding, or if it's determined to be in your best interest.

Additionally, your involvement may be stopped if your health deteriorates, if you become pregnant, if you choose not to continue with the research after being informed of any changes that may impact you, or if you fail to follow the study's guidelines. It's crucial to carefully consider these factors before deciding to participate in a clinical trial.

# Comparing Head and Neck Cancer Clinical Trials to Other Types

When it comes to clinical trials for head and neck cancer, participation is entirely optional, and you have the right to withdraw from the study at any time without any negative consequences.

If you're searching for <u>studies for head and neck cancer</u> from all over the world, you can go to clinicaltrials.gov, a website operated by the National Institutes of Health (NIH) that provides a comprehensive database of trials. You may narrow down your search by applying different criteria, such as location and medical condition.

In addition, Power's reference page has a list of active <u>head and neck clinical trials</u> that are presently recruiting participants.

### Online Resources for Understanding Clinical Trial Diversity

For individuals interested in learning more about clinical trial diversity, there are numerous online resources available. Here are a couple of articles that may be of interest to you:

Hurwitz, Brian. "Form and representation in clinical case reports." *Literature and Medicine* 25, no. 2 (2006): 216-240.

Bird, Chloe E. "Women's representation as subjects in clinical studies: a pilot study of research published in JAMA in 1990 and 1992." Women and health research: Ethical and legal issues of including women in clinical studies 2 (1994): 151-173.

These websites offer valuable information on the challenges surrounding clinical trial diversity and the proposed solutions.

# Ensuring Confidentiality in Research Studies

We take the privacy of the personal information collected for this research project very seriously. While we cannot guarantee that your personal information will remain completely confidential at all times, we have taken every possible measure to protect it. Please note that in some situations, it may be legally required to disclose your personal

information. However, we assure you that no research publications or presentations will contain your name or any other personally identifying information.

Your medical information may be accessed by a range of organizations, including accrediting bodies, government, and regulatory authorities (such as the FDA and OHRP), safety monitors, study sponsors, and authorized sponsor representatives, for research, quality assurance, and data analysis purposes.

On rare occasions, we may ask you to complete an "Authorization Form" outlining how we can use your information and with whom we may share it for this study.

Before sharing any of the information or research samples you provided for this study with Power researchers, researchers from other university institutions, or researchers from outside commercial firms for future research, we will first obtain your explicit consent. You can be assured that your confidential data will be removed and kept secure.

# Informed Consent Agreement

By signing this consent agreement, you acknowledge and agree to the following:

- You have read and fully understood this informed consent form. Before making a
  decision, you are encouraged to discuss this information with others and seek
  alternative viewpoints.
- You have received satisfactory answers to all of your questions about the research project and its methods, as well as all the information you need to participate in the study.
- You have considered the potential benefits, drawbacks, and alternatives to participating in the research.
- Your voluntary participation in the research study will not affect your ability to exercise your legal rights.
- You will be informed of any significant updates to the research study that may impact your decision to continue participating.
- This consent form has been provided to you and you have had the opportunity to ask any questions you may have.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Researcher's Signature | | |
| As the researcher, I ensured that th received a comprehensive explana participation is voluntary and fully in | tion of the study. I have also co | • |
| Signature of Researcher Who | Received Consent | |
| Name of Investigator | Signature of Investigator | Date |